CLINICAL TRIAL: NCT06627192
Title: Effect of Non-surgical Periodontal Therapy in Hypertensive Patients With Assessment of Endocan and TNF-a Levels in Gingival Crevicular Fluid (Case Control Study)
Brief Title: Effect of Non-surgical Periodontal Therapy in Hypertensive Patients With Assessment of Endocan and TNF-α Levels in GCF
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lana Nabil, Master's candidate, Ain Shams University
Other Study IDs: FDASU-RECD 1293 1123 1234
Record Dates: First submitted 2024-08-26; First posted 2024-10-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis; Hypertension; TNF Alpha; Endocan; GCF
Keywords: Peridontitis; Stage 2; Hypertension; Pro-inflammatory cytokines; GCF; NSPT; ELISA; Endocan; ESM-1; Biochemical assessment; Non-surgical periodontal therapy
MeSH Terms: conditions — Periodontitis; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 Case: Group Case (I):
  This group will include 20 patients diagnosed with stage II periodontitis and controlled hypertension. They will receive NSPT and oral hygiene measures will be instructed following treatment.
  Interventions: Procedure: NSPT, clinical and biochemical assesment
- Group 2 Control: This group will include 20 patients diagnosed with stage II periodontitis and no hypertension. They will receive NSPT and oral hygiene measures will be instructed following treatment.
  Interventions: Procedure: NSPT, clinical and biochemical assesment

INTERVENTIONS:
Procedure: NSPT, clinical and biochemical assesment — Biochemical assessment using ELISA kit for Endcan and TNF alpha GCF sample
  Other Names: ELISA kit for GCF sample test

SUMMARY:
There is a strong crossway relationship between periodontitis and hypertension. Hypertension is the most prevalent of cardiovascular diseases and its prevalence is increased by the presence of periodontitis. Periodontal attachment loss is higher in hypertension patients when compared to healthy subjects. Both are examples of non-communicable diseases (NCDs), also known as chronic inflammatory diseases, they tend to be of long duration and are the result of a combination of genetic, physiological and environmental factors. The lack of an appropriate balance between these factors results in cellular changes as well as the levels of cytokines with subsequent changes in clinical manifestations of periodontal diseases. Both periodontitis and hypertension are associated with inflammation and an increase in specific proinflammatory cytokines.

Aim of the study: To investigate the correlation between the clinical parameters and the levels of Endocan and TNF-α in gingival crevicular fluid (GCF) before and after non-surgical periodontal therapy (NSPT) in stage II periodontitis patients with hypertension in comparison to non-hypertensive patients.

DETAILED DESCRIPTION:
Clinical assessment of specific clinical parameters: plaque index, gingival index, probing depth, clinical attachment level (CAL) as primary outcome. Biochemical assessment of Endocan and TNF-α levels in GCF by Enzyme Linked Immunosorbent Assay (ELISA) as well as measurement of blood pressure at baseline and after 3 months as secondary outcomes.

Study procedures:

Details of the interventions, testing and follow up:

Group Case (I):

This group will include 20 patients diagnosed with stage II periodontitis and controlled hypertension. They will receive NSPT and oral hygiene measures will be instructed following treatment.

Group Control (II):

This group will include 20 patients diagnosed with stage II periodontitis and no hypertension. They will receive NSPT and oral hygiene measures will be instructed following treatment.

Study protocol and surgical steps:

Before enrollment, a detailed case history will be recorded. A calibrated standard aneroid sphygmomanometer. The average of 3 blood pressure values (systolic blood pressure SBP and diastolic blood pressure DBP), will be taken at 1 minute interval, this will be used in data analyses.

For all patients who are suitable for the study the following clinical evaluation parameters will be measured:

Plaque index (PI) Gingival index (GI) Probing depth (PD) Bleeding on probing (BOP) Clinical attachment level (CAL) Standardized periapical radiograph.

Note: Full mouth assessment will be done and then the deepest site will be evaluated for the GCF sample.

Baseline GCF samples will be taken the day after patients were clinically evaluated to prevent contamination with blood related to the probing of inflamed areas.

The sample areas will be insulated with cotton rolls to prevent saliva contamination and all supragingival plaque will be eliminated. The paper strips will be placed into the periodontal pocket and then permitted to remain for 30 seconds.

All patients will undergo full mouth NSPT, this will be done using ultrasonic and hand instruments.

The patients will receive oral hygiene instructions including tooth brushing using modified bass technique. All patients will be provided with toothbrush (soft), toothpaste (signal) and interdental cleaning with dental floss or interdental brush.

Two weeks follow-up to ensure that appropriate oral hygiene instructions are followed. The clinical parameter to be assessed will be PI and BOP, patients with PI 2 and BOP > 10% will be eliminated from the study.

Then clinical evaluation, collection of samples and measuring of SBP and DBP will be performed at 3 months after NSPT in both groups.

The Outcomes Assessment:

Clinical assessment. Biochemical assessment. Blood pressure measurement.

For clinical assessment the following clinical parameters including PI, GI, PD, BOP and CAL will be recorded for each individual at 1 site at baseline and 3 months postoperatively. Clinical parameters of PI and BOP will be assessed at 2 weeks, 4 weeks and 6 weeks follow ups to ensure proper oral hygiene. Regarding biochemical analysis, GCF samples will be collected preoperative and 3 months after NSPT. Blood pressure measurements will be taken before and after 3 months of NSPT.

Clinical Assessment The following clinical parameters will be taken using UNC15 Probe at baseline and 3 months postoperative.

Plaque index:

* no plaque.
* plaque recognized only by running a probe across the tooth surface.
* plaque visible to the naked eye.
* abundance of soft matter.

Gingival index:

* Normal gingiva
* Mild inflammation - slight edema. No bleeding on probing
* Moderate inflammation -redness, edema and glazing. Bleeding on probing.
* Severe inflammation - marked redness and edema. Ulceration. Tendency for spontaneous bleeding

Probing depth :

Will be measured from the gingival margin to the depth of the pocket at four points (mesio-facial, mid-facial, disto-facial and mid-lingual) to the nearest millimeter using UNC-15 periodontal probe. The average of the three facial points will be recorded as the facial probing depth (FPD) while the mid-lingual point will be recorded as the lingual probing depth.

Clinical attachment level (CAL):Will be measured from the CEJ to the depth of the periodontal pocket.

b) Biochemical Assessment:

Biochemical assessment will be done at the deepest pocket at baseline and 3 months after non-surgical periodontal therapy. Endocan and TNF-α levels will be determined using commercial human Endocan (ESM-1) and TNF-α ELISA Kits. Measurements will be performed according to the manufacturer's instructions.

c) Blood Pressure measurement: Systolic and diastolic Blood pressure measurement will be done according to, 2020 International Society of Hypertension Global Hypertension Practice Guidelines.

IX. Statistical Analysis The obtained results will be collected, tabulated, and subjected to appropriate statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II periodontitis and controlled hypertension (self-reported history of a diagnosis of HTN by a physician and blood pressure (SBP < 140 and DBP < 90).
* Both genders aged from 30-70.
* Minimum 20 natural teeth excluding third molars.
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow-up and maintenance program.

Exclusion Criteria:

* Smokers.
* Pregnant and lactating females.
* Patients with other systemic diseases, such as diabetes mellitus, rheumatoid arthritis and cancer.

(According to Cornell Medical Index-Health Questionnaire).

* Patients taking antibiotic, anti-inflammatory, and immunosuppressive therapy during the preceding 3 months before the start of the trial and during the study.
* Patients who have undergone any periodontal therapy in the last 6 months.

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stage II periodontitis and controlled hypertension (self-reported history of a diagnosis of HTN by a physician and blood pressure (SBP < 140 and DBP < 90).
  Both genders aged from 30-70. Minimum 20 natural teeth excluding third molars. Good compliance with the plaque control instructions following initial therapy. Availability for follow-up and maintenance program.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of PI plaque index | 3 months
  For clinical assessment the following clinical parameter PI plaque index will be recorded for each individual at 1 site at baseline and 3 months postoperatively. Clinical parameters of PI will be assessed at 2 weeks, 4 weeks and 6 weeks follow ups to ensure proper oral hygiene. Regarding biochemical analysis, GCF samples will be collected preoperative and 3 months after NSPT.
  Plaque index at deepest pocket will be measured.
Clinical assessment of BOP bleeding on probing | 3 months
  For clinical assessment the following clinical parameter BOP will be recorded for each individual at 1 site at baseline and 3 months postoperatively. Clinical parameters of BOP will be assessed at 2 weeks, 4 weeks and 6 weeks follow ups to ensure proper oral hygiene. Regarding biochemical analysis, GCF samples will be collected preoperative and 3 months after NSPT.
  bleeding on probing at deepest pocket will be measured
Clinical assessment of CAL clinical attachment loss | 3 months
  For clinical assessment the following clinical parameter CAL will be recorded.for each individual at 1 site at baseline and 3 months postoperatively. Regarding biochemical analysis, GCF samples will be collected preoperative and 3 months after NSPT.
  clinical attachment loss at deepest pocket will be recorded.
Clinical assessment of PD probing depth | 3 months
  For clinical assessment the following clinical parameter PD will be recorded for each individual at 1 site at baseline and 3 months postoperatively. Regarding biochemical analysis, GCF samples will be collected preoperative and 3 months after NSPT. PD at deepest pocket will be recorded.

SECONDARY OUTCOMES:
Biochemical assesment of Endocan | 3 months
  Using GCF samples and asses Endocan by ELISA kit
Biochemical assesment of TNF-α | 3 months
  Using GCF samples and asses TNF-α by ELISA kit

OTHER OUTCOMES:
Blood pressure measurement | 3 months
  Measure Systolic and dyastolic Blood pressure at baseline and at followup

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT06627192/Prot_002.pdf
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT06627192/ICF_003.pdf